CLINICAL TRIAL: NCT06678919
Title: AGMT Metastatic Colorectal Cancer Registry (mCRC) Third Line and Beyond
Status: Recruiting | Type: Observational
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Other Study IDs: AGMT_mCRC_3L and beyond-Reg
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: colorectal
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The Lymphoma registry will be accompanied by an optional biobanking program. Sample collection will be limited to patients that have signed an additional biobanking IC. The samples are taken as part of the clinical routine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Colorectal cancer (CRC) is the second leading cause of cancer-related death in the United States and Europe. Although selected patients with oligometastatic CRC undergo systemic therapy and surgery/local ablative therapy in curative intent, the treatment approach for the majority of metastatic CRC (mCRC) patients remains palliative with a median overall survival (OS) ranging between 9-38 months depending on various prognostic and predictive factors. Particularly in advanced stages (in the third line of therapy and beyond), interesting and promising results have recently been achieved with various treatment approaches. The aim of this registry is to establish a disease-specific registry to evaluate the treatment landscape of patients with mCRC who have already received at least two lines of therapy.

DETAILED DESCRIPTION:
This registry aims at retrospectively and prospectively evaluating the treatment landscape and clinical outcome of mCRC ≥3L in a collective attempt by including multiple oncologic centers in Austria.

Patient medical, testing and treatment information will be obtained through extraction of data from existing patient medical charts. Longitudinal follow-up data, including survival and tumor progression, will also be extracted from patient medical charts. Imaging studies ≥3L will be centrally collected in a virtual "imaging-bank" and tumor tissue samples of deceased patients will be stored in a central "bio-bank". Additionally, further biomaterial (e.g. ctDNA samples or DNA from DPYD genotyping) may be requested from the centres in case of specific research questions. The patient follow-up data will be obtained until patient death or loss to follow-up.

For documentation in the registry, no further diagnostic or therapeutic measures are required than those already necessary in general. Participation in the registry must not interfere with treatment routines. Only routine data, which have already been recorded in the patients' medical charts, is transferred to the electronic Case Report Forms. To maintain patient confidentiality, each patient will be assigned a unique patient identifying number upon enrollment; this number will accompany the patients' medical and other registry information throughout the lifetime of the registry.

A written consent must be obtained prior to the input of data. No informed consent is required from deceased patients.

Data will be collected from all sites willing to participate.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years with tissue-based diagnosis of mCRC
* ≥ 2 prior lines of palliative systemic therapy including 5-FU, irinotecan, oxaliplatin, anti-VEGF, anti-EGFR (in case of RAS/BRAF wildtype), anti-PD1- therapy (in case of MSI/MMRd) . (Exception: Patients who have received mFOLFOXIRI +/- anti-VEGF or anti- EGFR- 1L therapy or patients with ineligibility to receive 5-FU, oxaliplatin or irinotecan can be included after 1st line.)

Exclusion Criteria:

* Due to the non-interventional design of this registry, there are no specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interested sites that treat patients in this indication will be invited to participate in this registry
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 10 years
  Overall survival with the respective treatment protocols ≥3L
Progression free survival | 10 years
  Progression-free survival (PFS) with the respective treatments protocols ≥3L
Overall response rate (ORR) | 10 years
  Overall response rate (ORR) with the respective ≥3L treatment protocols
Blinded Independent Central Review (BICR) | 10 years
  Blinded Independent Central Review (BICR) based on the virtual imaging-bank
Identification of predictive biomarkers | 10 years
  Identification of predictive biomarkers for mCRC patient sub-cohorts of interest based on the centrally-located bio-bank

CONTACTS AND LOCATIONS:
Locations (7):
- Austria (7):
  - Ordensklinikum Linz, BHS - Interne I, Linz
  - KUK Linz - Med Campus III.: Univ.-Klinik für Hämatologie und Internistische Onkologie, Linz
  - LKH Feldkirch: Innere Medizin II/ Interne E (Hämatologie und Onkologie), Rankweil
  - Department of Internal Medicine III, Paracelsus Medical University Salzburg, Salzburg
  - Klinikum Steyr: Innere Medizin II: Onkologie, Gastroenterologie, Angiologie, Steyr
  - Klinikum Wels: Abteilung für Innere Medizin IV, Wels
  - KH Zams: Innere Medizin Internistische Onkologie und Hämatologie, Zams